CLINICAL TRIAL: NCT01894230
Title: Genetically Guided Statin Therapy to Improve Medication Adherence
Brief Title: Genetically Guided Statin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00044989; Pro00045542 (Other: DUHS IRB)
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Hypercholesterolemia; Hydroxy-methylglutaryl-coenzyme A (HMG Co-A) Reductase Inhibitors Adverse Reaction
Keywords: high cholesterol; genetic testing; medication adherence; statins; Adverse Effects; pharmacogenetics
MeSH Terms: conditions — Hypercholesterolemia; Medication Adherence | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Genotype results plus usual care (Experimental): SLCO1B1*5 allele testing, results reported at randomization: genetic testing for SLCO1B1*5 allele and reporting of results to patient and provider at randomization.
  Interventions: Genetic: SLCO1B1*5 allele testing, results reported at randomization; Genetic: Genetic testing for SLCO1B1*5 allele
- Usual care only (Active Comparator): SLCO1B1*5 allele testing, results reported at end of study: genetic testing for SLCO1B1*5 allele and reporting of results to patient and provider at end of study
  Interventions: Genetic: SLCO1B1*5 allele testing, results reported at end of study; Genetic: Genetic testing for SLCO1B1*5 allele

INTERVENTIONS:
Genetic: SLCO1B1*5 allele testing, results reported at randomization — Genetic testing for SLCO1B1*5 allele and reporting of results to patient and provider at randomization
  Other Names: genotype informed statin therapy (GIST)
  Arms: Genotype results plus usual care
Genetic: SLCO1B1*5 allele testing, results reported at end of study — Genetic testing for SLCO1B1*5 allele and reporting of results to patient and provider at end of study
  Arms: Usual care only
Genetic: Genetic testing for SLCO1B1*5 allele — Blood test for SLCO1B1*5 allele

SUMMARY:
The purpose of this study is to examine if using genetics can improve statin adherence in patients who should be taking statins but are not because of prior side effects. This study will assist physicians/providers in making a personalized health care plan for prevention of cardiovascular disease.

DETAILED DESCRIPTION:
Hydroxy-methylglutaryl-coenzyme A (HMG Co-A) reductase inhibitors ("statins") are commonly prescribed to lower low density lipoprotein cholesterol (LDLc) and to prevent cardiovascular disease (CVD), a leading cause of morbidity and mortality. Long-term adherence to statins in the primary care environment is challenging; consequences of statin non-adherence include higher LDLc levels, hospitalizations, costs, and death due to CVD.

Medication non-adherence is complex and multifactorial and can be associated with a number of factors including medication cost, complexity of medication regimen, poor provider-patient relationship / communication, and adverse side effects. For statins, side effects such as muscle aches, cramping, and pain (referred to broadly as statin-related myopathy) are a frequent cause of non-adherence. These symptoms are non-specific and are frequent reasons for stopping statin therapy, due to patient or provider concern about the possibility of statin-related myopathy. Many patients may be needlessly deprived of the cardiovascular benefits of long-term statin use.

A genetic risk factor for statin myopathy and subsequent non-adherence has recently been identified. In a genome-wide association study, a genetic variant (named SLCO1B1*5) was a main contributor of statin myopathy. It was demonstrated that the SLCO1B1*5 variant is not only a predictor of myopathy, but also of premature statin discontinuation. The risk with the *5 allele is statin specific: greatest with simvastatin and atorvastatin use, the least with pravastatin or rosuvastatin. Therefore, the SLCO1B1*5 variant is common, can predict myopathy, subsequent non-adherence, and due to its statin-specific effects creates a novel research paradigm for personalizing statins to an individual's genetic profile. Carriers of the SLCO1B1*5 variant may do best on rosuvastatin, pravastatin, or fluvastatin whereas non-carriers may be treated with any statin.

The objective of this study is to conduct a randomized trial comparing two strategies:

1. genetically guided statin therapy vs.
2. usual care (i.e., a strategy without genetics) on the effects of statin adherence and LDLc lowering.

The overall hypothesis is that genetically guided statin therapy will lead to greater statin adherence and lower LDLc when compared to a non-guided strategy. The design of this trial will randomize primary care patients within Duke University Health System (DUHS) and travis Air Force Base (TAFB) clinics that are nonadherent to statins due to prior side-effects in an unblinded, 1:1 fashion, stratified by SLCO1B1*5 genotype.

ELIGIBILITY:
Inclusion Criteria:

* Current patient (defined as seen in the last year) of the Duke Primary Care at Pickett Road, Pickens Family Medicine Center or Travis Air Force Base
* Age greater than or equal to 18 years
* Current non-utilization of statin therapy for either of the following reasons: (a) Prior side effects thought to be attributed by the patient to statin use AND/OR (b) Physician removal of statin due to presumed associated side effects
* No statin use for the past 6 weeks
* Active email account
* Computer access available in order to complete on-line surveys
* Ability to provide informed consent

Exclusion Criteria:

* Prior rhabdomyolysis, or Creatine Kinase (CK) elevation > 10 times the upper limit of normal with any statin therapy
* Prior unexplained elevation in hepatic enzymes [Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) > 3 times upper limit of normal] with any statin therapy
* Current daily grapefruit juice usage (on average >1quart/day)
* Expected long term use (longer than 3 months) of the following medications known to interfere with statin metabolism or disposition at time of enrollment until the randomization is complete. However, short-term (<14 days) is allowed for the duration of the study
* Participation in a drug research study in the past 30 days
* Previous use of 4 or more statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2013-07; Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Voora, MD, Principal Investigator — Duke University; Henry Lau, MD, Principal Investigator — David Grant US Air Force Medical Center
Locations (2):
- United States (2):
  - David Grant US Air Force Medical Center, Travis Air Force Base, California
  - Duke University, Durham, North Carolina

REFERENCES:
- [Derived] Peyser B, Perry EP, Singh K, Gill RD, Mehan MR, Haga SB, Musty MD, Milazzo NA, Savard D, Li YJ, Trujilio G, Voora D. Effects of Delivering SLCO1B1 Pharmacogenetic Information in Randomized Trial and Observational Settings. Circ Genom Precis Med. 2018 Sep;11(9):e002228. doi: 10.1161/CIRCGEN.118.002228. PMID 30354330
- [Derived] Ramsey LB, Johnson SG, Caudle KE, Haidar CE, Voora D, Wilke RA, Maxwell WD, McLeod HL, Krauss RM, Roden DM, Feng Q, Cooper-DeHoff RM, Gong L, Klein TE, Wadelius M, Niemi M. The clinical pharmacogenetics implementation consortium guideline for SLCO1B1 and simvastatin-induced myopathy: 2014 update. Clin Pharmacol Ther. 2014 Oct;96(4):423-8. doi: 10.1038/clpt.2014.125. Epub 2014 Jun 11. PMID 24918167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight participants that signed a consent either withdrew consent, were lost-to follow up, or were screen-failures and thus were not randomized.
Groups:
- Genotype Results Plus Usual Care: * Genetic testing for SLCO1B1*5 allele
  * Reporting for SLCO1B1*5 allele at randomization
  Reporting for SLCO1B1*5 allele at randomization: Reporting of genetic test results to patient and provider at randomization
  Genetic testing for SLCO1B1*5 allele: Blood test for SLCO1B1*5 allele
- Usual Care Only: * Genetic testing for SLCO1B1*5 allele
  * Reporting for SLCO1B1*5 allele at the end of study
  Reporting for SLCO1B1*5 allele at the end: Usual care recommendations provided to patient and provider at randomization. Genotyping results provided at the end of study.
  Genetic testing for SLCO1B1*5 allele: Blood test for SLCO1B1*5 allele
Period: Overall Study
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
Started | 83 | 76
Completed | 76 | 69
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Non-adherent | 0 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only | Total
Number analyzed (Participants) | 83 | 76 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.2) | 62.5 (11.5) | 62.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 50 | 91
  Male | 42 | 26 | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 66 | 61 | 127
  Race/Ethnicity: Black/African American | 14 | 11 | 25
  Race/Ethnicity: Other | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 83 | 76 | 159

OUTCOME MEASURES:

1. Primary Outcome: Morisky Medication Adherence Scale (MMAS) Score
Description: The Morisky Medication Adherence Scale (MMAS) is a self-reported measure of adherence, collected at baseline for general medication and at 3 and 8 months of followup for statin specific adherence. The eight-item MMAS survey will be used. This is a modified version of the original four-item MMAS capturing further aspects of adherence behavior. The survey includes 8 yes/no items that are summed to create an overall adherence score ranging from of 0 to 8, with higher scores indicating better adherence. The primary hypothesis is that the genetically guided statin therapy leads to greater adherence of statin therapy, corresponding to a higher MMAS score.
Time Frame: 3 months and 8 months
Population: Only participants who re-initiated statin use were eligible to do statin specific MMAS and included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Genotype Results Plus Usual Care: -Genetic testing for SLCO1B1*5 allele reported to patient and provider at randomization
- Usual Care Only: -Genetic testing for SLCO1B1*5 allele reported to patient and provider at the end of study
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
Number analyzed (Participants) | 37 | 25
units on a scale
  MMAS Score 3 Months | 6.8 (1.5) | 6.9 (1.6)
  MMAS Score 8 Months: number analyzed (Participants) | 28 | 22
  MMAS Score 8 Months | 6.8 (1.7) | 7.1 (1.3)
Statistical Analysis 1: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 3; p = 0.96, Regression, Linear; Slope = -0.0189, Standard Error of Mean 0.3986
Statistical Analysis 2: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 8; p = 0.57, Regression, Linear; Slope = -0.2468, Standard Error of Mean 0.4315

2. Secondary Outcome: Low Density Lipoprotein Cholesterol (LDLc) at Baseline, Month 3 and Month 8
Description: The continuous outcomes LDLc will be modeled as a linear regression with arm and baseline LDL as predictors.
Time Frame: Baseline, Month 3, Month 8
Population: All subjects with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
Number analyzed (Participants) | 83 | 76
mg/dL
  Baseline LDLc | 152.7 (41.1) | 157.6 (41.9)
  Month 3 LDLc: number analyzed (Participants) | 78 | 70
  Month 3 LDLc | 131.9 (42) | 144.4 (43)
  Month 8 LDLc: number analyzed (Participants) | 59 | 60
  Month 8 LDLc | 128.6 (37.9) | 141 (44.4)
Statistical Analysis 1: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 3; p = 0.0482, Regression, Linear; Slope = -11.32, Standard Error of Mean 5.68
Statistical Analysis 2: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 8; p = 0.12, Regression, Linear; Slope = -9.9, Standard Error of Mean 6.333

3. Secondary Outcome: Medication Possession Ratio (MPR) From Baseline to Last Patient Follow-up
Description: Medication possession ratio will be calculated based on number of statin medication refills over time from randomization to end of follow up. MPR is calculated as follows: 1.Sum of the days' supply of all statin medications is the sum of the number of pills dispensed for each statin prescription during follow up (taken from 3-month, 4-month and 8-month statin utilization review) 2.Sum of the days of follow up = date of 8-month follow up survey - date of randomization 3.MPR = #1/#2 MPR will be modeled as a linear regression with arm, genotype, and site as predictors.
Time Frame: Baseline to Last patient follow-up in study (3 months or 8 months)
Population: Only subjects who re-initiated statin medication and reported statin medication refills were included in the analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
Number analyzed (Participants) | 24 | 20
ratio | 0.632 (0.333) | 0.685 (0.483)
Statistical Analysis 1: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — MPR calculated from baseline to last patient follow-up (3 months or 8 months); p = 0.6692, Regression, Linear; Slope = -0.053, Standard Error of Mean 0.091

4. Secondary Outcome: Number of Participants Reporting New Statin Prescriptions
Description: The number of new prescriptions is binary and will be modeled with logistic regression with arm, genotype, and site as predictors. Any variables imbalanced between arms will also be included as covariates.
Time Frame: Baseline, Month 3, Month 8
Population: Only subjects reporting new prescriptions were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
Number analyzed (Participants) | 74 | 71
Participants
  Baseline to Month 3 | 41 | 27
  Month 3 to Month 8: number analyzed (Participants) | 56 | 62
  Month 3 to Month 8 | 4 | 4
Statistical Analysis 1: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Baseline to Month 3; p = 0.0371, Regression, Logistic; Odds Ratio (OR) = 2.025, 95% CI 2-sided [1.043 to 3.929]
Statistical Analysis 2: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 3 to Month 8; p = 0.8815, Regression, Logistic; Odds Ratio (OR) = 1.115, 95% CI 2-sided [0.265 to 4.687]

5. Secondary Outcome: Brief Pain Inventory (BPI) Score - Pain Severity at Month 3 and Month 8
Description: Brief Pain Inventory data will be taken from 3 and 8-month follow up Patient Surveys. Pain severity and pain interference will be compared between groups. Both of these measures will be modeled as a linear regression with arm, genotype, and site as predictors. Transformations of the response may be explored depending on the distribution of the regression residuals. Baseline pain scores will also be included as a covariate to account for baseline variability.
  Scores range from 0-10. Higher scores indicate higher pain severity.
Time Frame: Month 3 and Month 8
Population: Only subjects that completed the Brief Pain Inventory surveys were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
Number analyzed (Participants) | 74 | 67
units on a scale
  Month 3 | 1.608 (1.978) | 1.493 (1.854)
  Month 8: number analyzed (Participants) | 49 | 61
  Month 8 | 1.939 (1.93) | 1.689 (2.248)
Statistical Analysis 1: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 3; p = 0.5965, Regression, Linear; Slope = 0.143, Standard Error of Mean 0.270
Statistical Analysis 2: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 8; p = 0.4579, Regression, Linear; Slope = 0.258, Standard Error of Mean 0.346

6. Secondary Outcome: Brief Pain Inventory (BPI) Score - Pain Interference at Month 3 and Month 8
Description: Brief Pain Inventory data will be taken from 3 and 8-month follow up Patient Surveys. -Pain severity and pain interference will be compared between groups -Both of these measures will be modeled as a linear regression with arm as predictor. Baseline pain scores will also be included as a covariate to account for baseline variability.
  Scores range from 0-10. Higher scores indicate higher pain interference with daily activities.
Time Frame: Month 3 and Month 8
Population: Only subjects that completed the Brief Pain Inventory surveys were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
Number analyzed (Participants) | 74 | 70
units on a scale
  Month 3 | 2.108 (1.141) | 1.971 (1.049)
  Month 8: number analyzed (Participants) | 56 | 61
  Month 8 | 1.964 (0.894) | 1.689 (0.941)
Statistical Analysis 1: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 3; p = 0.5477, Regression, Linear; Slope = 0.098, Standard Error of Mean 0.163
Statistical Analysis 2: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 8; p = 0.0429, Regression, Linear; Slope = 0.298, Standard Error of Mean 0.145

7. Secondary Outcome: Change in Short Form -12 Item (SF-12) Health Survey - Physical Component (PC)
Description: Month 3 and Month 8 SF12 scores for mental and physical health will be compared. Both of these measures will be modeled as a linear regression with arm as predictor. Baseline SF-12 scores will also be included as a covariate to account for baseline variability.
  Ranges from 0 to 100, where a zero score indicates the lowest level of physical health measured by the scales and 100 indicates the highest level of physical health
Time Frame: Baseline, Month 3, Month 8
Population: Only subjects that completed the SF-12 Health Survey were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
Number analyzed (Participants) | 82 | 76
units on a scale
  Baseline | 42.244 (6.554) | 41.692 (7.281)
  Month 3: number analyzed (Participants) | 74 | 70
  Month 3 | 41.389 (6.891) | 41.566 (5.708)
  Month 8: number analyzed (Participants) | 56 | 61
  Month 8 | 42.179 (6.754) | 41.359 (5.721)
Statistical Analysis 1: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 3; p = 0.8106, Regression, Linear; Slope = -0.211, Standard Error of Mean 0.881
Statistical Analysis 2: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 8; p = 0.5233, Regression, Linear; Slope = 0.646, Standard Error of Mean 1.009

8. Secondary Outcome: Change in Short Form -12 Item (SF-12) Health Survey - Mental Component (MC)
Description: Month 3 and Month 8 SF12 scores for mental and physical health will be compared. Both of these measures will be modeled as a linear regression with arm as predictor. Baseline SF-12 scores will also be included as a covariate to account for baseline variability.
  Ranges from 0 to 100, where a zero score indicates the lowest level of mental health measured by the scales and 100 indicates the highest level of mental health.
Time Frame: Baseline, Month 3, Month 8
Population: Only subjects that completed the SF-12 Health Survey were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale 0 to 100
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
Number analyzed (Participants) | 82 | 76
units on a scale 0 to 100
  Baseline | 43.393 (11.801) | 44.101 (12.114)
  Month 3: number analyzed (Participants) | 74 | 70
  Month 3 | 42.835 (11.438) | 44.595 (11.361)
  Month 8: number analyzed (Participants) | 56 | 61
  Month 8 | 43.776 (11.344) | 44.327 (11.987)
Statistical Analysis 1: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 3; p = 0.6841, Regression, Linear; Slope = -0.6001, Standard Error of Mean 1.472
Statistical Analysis 2: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 8; p = 0.6658, Regression, Linear; Slope = -0.771, Standard Error of Mean 1.781

9. Secondary Outcome: Physical Activity Scale Score
Description: Activity levels will be compared at the end of 8-months. Activity levels are defined by a five-level ordinal variable (0-4; higher level corresponding to higher activity). which was calculated based on survey answers. An ordinal logistic regression model will be used with arm as predictor. The assumption of proportional odds will be checked, and if it is not met, a multinomial regression model will be used. -Baseline physical activity will also be included as a covariate to account for baseline variability.
  Scale score (0-4): 0 - Inactivity, 1 - Ligh-intensity activity, 2 - moderate-intensity activity, 3 - Hard-intensity activity, 5 - very hard-intensity activity
Time Frame: Baseline and Month 8
Population: Only subjects that completed the Physical Activity survey were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
Number analyzed (Participants) | 74 | 72
units on a scale
  Baseline | 1.838 (1.629) | 1.736 (0.822)
  Month 8: number analyzed (Participants) | 52 | 60
  Month 8 | 1.923 (1.152) | 1.667 (1.02)
Statistical Analysis 1: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 8; p = 0.8384, Regression, Logistic; Ordinal Logistic; Odds Ratio (OR) = 1.085, 95% CI 2-sided [0.495 to 2.380]

10. Secondary Outcome: Beliefs About Medications (BMQ) Score at Baseline, Month 3 and Month 8
Description: * Questionnaire administered at baseline, 3 months, and 8 months
  * This instrument assesses beliefs regarding necessity and concerns related to disease-specific medications
  * The score ranges from 5 to 25 representing the sum of 5 questions. This will be modeled with linear regression including treatment as predictor. Baseline BMQ scores will also be included as a covariate to account for baseline variability.
  Higher score corresponds to higher thought necessity and higher thought concerns about taking the medication. The higher the necessity score, the more the patient believed statins necessary for their health. The higher the concerns score, the more the patient was concerned about taking stains (side effects).
Time Frame: Baseline, Month 3, Month 8
Population: Only subjects that completed the Beliefs About Medications questionnaire were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
Number analyzed (Participants) | 82 | 75
units on a scale
  Baseline, BMQ Necessity | 13.878 (3.49) | 13.893 (3.443)
  Month 3, BMQ Necessity: number analyzed (Participants) | 72 | 65
  Month 3, BMQ Necessity | 14.347 (3.75) | 13.185 (3)
  Month 8, BMQ Necessity: number analyzed (Participants) | 54 | 60
  Month 8, BMQ Necessity | 14.148 (3.983) | 13.9 (3.487)
  Baseline, BMQ Concerns: number analyzed (Participants) | 79 | 75
  Baseline, BMQ Concerns | 15.962 (3.345) | 16.067 (2.974)
  Month 3, BMQ Concerns: number analyzed (Participants) | 70 | 63
  Month 3, BMQ Concerns | 14.471 (3.984) | 15.333 (3.914)
  Month 8, BMQ Concerns: number analyzed (Participants) | 53 | 59
  Month 8, BMQ Concerns | 13.585 (4.088) | 14.593 (3.71)
Statistical Analysis 1: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 3 BMQ Necessity; p = 0.0486, Regression, Linear; Slope = 1.163, Standard Error of Mean 0.584
Statistical Analysis 2: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 8, BMQ Necessity; p = 0.7235, Regression, Linear; Slope = 0.248, Standard Error of Mean 0.67
Statistical Analysis 3: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 3, BMQ Concerns; p = 0.2113, Regression, Linear; Slope = -0.862, Standard Error of Mean 0.686
Statistical Analysis 4: Comparison: Genotype Results Plus Usual Care vs Usual Care Only; Test type: Equivalence — Month 8, BMQ Concerns; p = 0.1739, Regression, Linear; Slope = -1.0083, Standard Error of Mean 0.737

ADVERSE EVENTS:
Time Frame: Baseline through Month 8
Arm/Group | Genotype Results Plus Usual Care | Usual Care Only
All-Cause Mortality (participants affected / at risk) | 1/83 | 0/76
Serious Adverse Events (participants affected / at risk) | 4/83 | 6/76
Other Adverse Events (participants affected / at risk) | 1/83 | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genotype Results Plus Usual Care (N=83) | Usual Care Only (N=76)
Liver function testing abnormality (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 2 (2)
Hospitalization for bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea, vomiting, abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Suspected MRSA bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genotype Results Plus Usual Care (N=83) | Usual Care Only (N=76)
Stroke (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes